CLINICAL TRIAL: NCT02120690
Title: Trigeminal Nerve Stimulation (TNS) as a Complementary Strategy in the Treatment of Fibromyalgia, Open Label Study
Brief Title: Trigeminal Nerve Stimulation (TNS) in the Treatment of Fibromyalgia
Acronym: TNS-FMA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Santa Casa Medical School (Other)
Responsible Party: Principal Investigator, Pedro Shiozawa, Coordinator - Laboratory of Clinical Neuromodualtion, Santa Casa Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNS-FMA
Record Dates: First submitted 2014-04-20; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Fibromyalgia
Keywords: pain; fibromyagia; TNS
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trigeminal nerve stimulation - active (Experimental): 10-day TNS interventional protocol over an 10-day follow-up
  Interventions: Device: Trigeminal nerve stimulation
- Trigeminal nerve stimulation (Sham Comparator): 10-day sham interventional protocol over an 10-day follow-up
  Interventions: Device: Trigeminal nerve stimulation

INTERVENTIONS:
Device: Trigeminal nerve stimulation — 10-day TNS interventional protocol over an 10-day follow-up. Subjects will have electrodes (Superior Silver 1.25-in. diameter) placed on their foreheads to stimulate the V1 branches of the trigeminal nerve bilaterally for approximately 30 minutes each day. Current was adjusted to maintain comfortable but perceptible levels of stimulation

SUMMARY:
To the investigators knowledge there are no studies of Trigeminal Nerve Stimulation (TNS) for fibromyalgia. TNS may modify overlapping mood and fibromyalgia pain regulation circuitry. The investigators hypothesized that patients with fibromyalgia might experience a clinically significant reduction in daily pain if investigators were to administer TNS in a manner similar to experimental antidepressant protocols.

ELIGIBILITY:
Inclusion Criteria:

* We will adopt the following inclusion criteria: (1) patients between 18 and 69 years; (2) patients with a diagnosis of fibromyalgia according to a trained phisycian; (3) score greater than or equal to 5 on the VAS for pain; (4) agreement to participate in the study as recommended in the IC.

Exclusion Criteria:

* Exclusion criteria we cite: (1) patients with psychiatric hospitalization indicated; (2) patients with psychiatric comorbidity; (3) patients with a diagnosis of personality disorder; (4) presence of severe neurological or medical diseases such as neoplasms in activity, neurodegenerative diseases and chronic decompensated.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
VAS for pain | 10 day-follow up
  Comparison between VAS for pain after intervention protocol and baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Shiozawa, MD, Study Director — Clinical Neuromodulation Laboratory - Santa Casa Medical School; Marcelo V Perez, MD, PhD, Principal Investigator — Department of Anestesiology - ISCMSP; Quirino Corderio, MD, PhD, Study Chair — Department of Psychiatry - ISCMSP
Locations (1):
- Centro de Atencao Integrada à Saúde Mental, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Collado A, Conesa A. [Pharmacologic treatment of fibromyalgia: Towards chemical neuromodulation]. Reumatol Clin. 2009 Aug;5 Suppl 2:27-31. doi: 10.1016/j.reuma.2009.04.003. Epub 2009 Jul 9. Spanish. PMID 21794655
- [Background] Tzabazis A, Aparici CM, Rowbotham MC, Schneider MB, Etkin A, Yeomans DC. Shaped magnetic field pulses by multi-coil repetitive transcranial magnetic stimulation (rTMS) differentially modulate anterior cingulate cortex responses and pain in volunteers and fibromyalgia patients. Mol Pain. 2013 Jul 2;9:33. doi: 10.1186/1744-8069-9-33. PMID 23819466
- [Background] Short BE, Borckardt JJ, Anderson BS, Frohman H, Beam W, Reeves ST, George MS. Ten sessions of adjunctive left prefrontal rTMS significantly reduces fibromyalgia pain: a randomized, controlled pilot study. Pain. 2011 Nov;152(11):2477-2484. doi: 10.1016/j.pain.2011.05.033. Epub 2011 Jul 20. PMID 21764215
- [Background] Ozgocmen S, Yoldas T, Kamanli A, Yildizhan H, Yigiter R, Ardicoglu O. Auditory P300 event related potentials and serotonin reuptake inhibitor treatment in patients with fibromyalgia. Ann Rheum Dis. 2003 Jun;62(6):551-5. doi: 10.1136/ard.62.6.551. PMID 12759293